CLINICAL TRIAL: NCT02902770
Title: A Randomized Trial Comparing the Combination of Intravenous Lidocaine and Ketorolac to Either Analgesics Alone for ED Patients With Acute Renal Colic
Brief Title: Intravenous Lidocaine and Ketorolac for Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-03-09
Record Dates: First submitted 2016-09-05; First posted 2016-09-16 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Pain
Keywords: Pain; Lidocaine; Ketorolac
MeSH Terms: conditions — Pain | interventions — Lidocaine; Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lidocaine and normal saline push (Active Comparator): 1.5mg/kg IV Lidocaine Drip (given over 10 minutes) and normal saline push
  Interventions: Drug: Lidocaine; Drug: Normal Saline Push
- Ketorolac and normal saline drip (Active Comparator): IV Ketorolac Tromethamine 30mg push and 10 minute normal saline drip
  Interventions: Drug: Ketorolac Tromethamine; Drug: Normal Saline Drip
- Lidocaine and Ketorolac (Active Comparator): IV Lidocaine Drip and IV Ketorolac Push
  Interventions: Drug: Lidocaine; Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Lidocaine — 1.5 mg/kg IV lidocaine drip (given over 10 minutes)
  Other Names: Xylocaine
  Arms: Lidocaine and Ketorolac; Lidocaine and normal saline push
Drug: Ketorolac Tromethamine — IV ketorolac 30mg push
  Other Names: Toradol
  Arms: Ketorolac and normal saline drip; Lidocaine and Ketorolac
Drug: Normal Saline Drip — Normal Saline Drip Placebo given over 10 minutes
  Other Names: Normal Saline
  Arms: Ketorolac and normal saline drip
Drug: Normal Saline Push — Normal Saline Push Placebo
  Other Names: Normal Saline
  Arms: Lidocaine and normal saline push

SUMMARY:
The literature regarding analgesic modalities, their combinations and routes of administrations for patients with pain related to renal colic is expanding. NSAID's (IV ketorolac) and opioids (morphine) constitutes the mainstay of treatment of renal colic either alone or in combinations. Despite their synergism and analgesic superiority when administered together, both classes of these medications possess a set of unfavorable side effects that limit their use. Emerging data of the use of IV lidocaine for patients with renal colic demonstrated good analgesic efficacy and safety profile. However, none of the trials directly compared lidocaine to ketorolac or the combination of both as viable options in patients unable to tolerate or to have serious contraindications to opioids. We designed a double-blinded, randomized, controlled trial to evaluate analgesic efficacy, safety and feasibility of non-opioid analgesics and their combinations in patients with renal colic. The hypothesis and proposed study will try to determine if a combination of IV lidocaine and reduced dose of IV ketorolac is superior to either drug alone and if this non-opioid analgesic modality is effective for controlling pain of renal colic origin.

DETAILED DESCRIPTION:
The investigators designed a double-blind, randomized, clinical trial to evaluate analgesic efficacy, safety and feasibility of non-opioid analgesics IV Lidocaine and IV Ketorolac and combination of both in patients with renal colic. The hypothesis and proposed study will try to determine if a combination of IV lidocaine and IV ketorolac is superior to either drug alone and if this non-opioid analgesic combination is effective for controlling pain of renal colic origin. The trial will compare pain scores at 15 min and 30 min between and within the three treatment groups of the study: IV ketorolac 30mg push and 10 minute normal saline drip placebo, 1.5mg/kg IV lidocaine drip (given over 10 minutes) and normal saline push placebo, or IV ketorolac push and IV lidocaine drip.

Once a patient is enrolled, the on duty ED pharmacist will prepare any one of the three treatment groups based on a predetermined randomization list generated via SPSS 19.0.The study investigators will record pain scores, vital signs, and side effects at baseline, 15, 30 and 60 minutes post-medication administration. If the patient still reports pain of five or greater and requests additional pain relief then morphine at 0.1mg/kg will be given as the rescue analgesic. Blinding of medication from the patient, research team, and staff will be strictly maintained by the pharmacist investigators.

Sample Size Calculation:

Fifty per group or 150 is needed given a standard 1.3 as the minimum clinically significant score and 3.0 as our standard deviation at 80% power and a=.05.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine Patient
* clinical diagnosis of acute renal colic
* pain score of >=5 out of 10 on the numeric rating scale
* - age 18 - 64 years of age

Exclusion Criteria:

* documented or suspected pregnancy, breastfeeding
* contraindication to nonsteroidal anti-inflammatory drugs or lidocaine
* known renal dysfunction
* received analgesics within 4 hours before presentation
* history of bleeding diathesis
* history of peptic ulcer disease
* current use of warfarin
* HR<50 or >150
* history of cardiac arrhythmias
* peritonitis or presence of any peritoneal sign
* altered mental status
* weight > 100kg

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10-04 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golzari SE, Soleimanpour H, Rahmani F, Zamani Mehr N, Safari S, Heshmat Y, Ebrahimi Bakhtavar H. Therapeutic approaches for renal colic in the emergency department: a review article. Anesth Pain Med. 2014 Feb 13;4(1):e16222. doi: 10.5812/aapm.16222. eCollection 2014 Feb. PMID 24701420
- [Background] Talati, J, Tiselius, H.-G, Albala, D.M, YE, Z. Urolithiasis: Basic Science and Clinical Practice. Springer Science & Business Media, Dec 22, 2012
- [Background] Sandhu DP, Iacovou JW, Fletcher MS, Kaisary AV, Philip NH, Arkell DG. A comparison of intramuscular ketorolac and pethidine in the alleviation of renal colic. Br J Urol. 1994 Dec;74(6):690-3. doi: 10.1111/j.1464-410x.1994.tb07107.x. PMID 7827834
- [Background] Larkin GL, Peacock WF 4th, Pearl SM, Blair GA, D'Amico F. Efficacy of ketorolac tromethamine versus meperidine in the ED treatment of acute renal colic. Am J Emerg Med. 1999 Jan;17(1):6-10. doi: 10.1016/s0735-6757(99)90003-7. PMID 9928687
- [Background] O'Connor A, Schug SA, Cardwell H. A comparison of the efficacy and safety of morphine and pethidine as analgesia for suspected renal colic in the emergency setting. J Accid Emerg Med. 2000 Jul;17(4):261-4. doi: 10.1136/emj.17.4.261. PMID 10921813
- [Background] Safdar B, Degutis LC, Landry K, Vedere SR, Moscovitz HC, D'Onofrio G. Intravenous morphine plus ketorolac is superior to either drug alone for treatment of acute renal colic. Ann Emerg Med. 2006 Aug;48(2):173-81, 181.e1. doi: 10.1016/j.annemergmed.2006.03.013. PMID 16953530
- [Background] Catapano MS. The analgesic efficacy of ketorolac for acute pain. J Emerg Med. 1996 Jan-Feb;14(1):67-75. doi: 10.1016/0736-4679(95)02052-7. PMID 8655940
- [Background] Castellsague J, Riera-Guardia N, Calingaert B, Varas-Lorenzo C, Fourrier-Reglat A, Nicotra F, Sturkenboom M, Perez-Gutthann S; Safety of Non-Steroidal Anti-Inflammatory Drugs (SOS) Project. Individual NSAIDs and upper gastrointestinal complications: a systematic review and meta-analysis of observational studies (the SOS project). Drug Saf. 2012 Dec 1;35(12):1127-46. doi: 10.2165/11633470-000000000-00000. PMID 23137151
- [Background] Duthie DJ, Nimmo WS. Adverse effects of opioid analgesic drugs. Br J Anaesth. 1987 Jan;59(1):61-77. doi: 10.1093/bja/59.1.61. PMID 2881564
- [Background] Soleimanpour H, Hassanzadeh K, Mohammadi DA, Vaezi H, Esfanjani RM. Parenteral lidocaine for treatment of intractable renal colic: a case series. J Med Case Rep. 2011 Jun 29;5:256. doi: 10.1186/1752-1947-5-256. PMID 21714904
- [Background] Soleimanpour H, Hassanzadeh K, Vaezi H, Golzari SE, Esfanjani RM, Soleimanpour M. Effectiveness of intravenous lidocaine versus intravenous morphine for patients with renal colic in the emergency department. BMC Urol. 2012 May 4;12:13. doi: 10.1186/1471-2490-12-13. PMID 22559856
- [Derived] Motov S, Fassassi C, Drapkin J, Butt M, Hossain R, Likourezos A, Monfort R, Brady J, Rothberger N, Mann SS, Flom P, Gulati V, Marshall J. Comparison of intravenous lidocaine/ketorolac combination to either analgesic alone for suspected renal colic pain in the ED. Am J Emerg Med. 2020 Feb;38(2):165-172. doi: 10.1016/j.ajem.2019.01.048. Epub 2019 Jan 30. PMID 30770244

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine and Normal Saline Push | Ketorolac and Normal Saline Drip | Lidocaine and Ketorolac
Started | 50 | 50 | 50
Completed | 50 | 50 | 50
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine and Normal Saline Push | Ketorolac and Normal Saline Drip | Lidocaine and Ketorolac | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (11.0) | 42.3 (10.5) | 41.9 (10.4) | 41.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 22 | 67
  Male | 27 | 28 | 28 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 30 Minutes
Description: The trial will compare the patient's pain score on a 11 point Likert scale, ranging from 0 to 10 with 0 being no pain, 5 moderate pain and 10 very severe pain, at 30 minutes
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine and Normal Saline Push | Ketorolac and Normal Saline Drip | Lidocaine and Ketorolac
Number analyzed (Participants) | 50 | 50 | 50
score on a scale | 5.52 (3.07) | 3.88 (2.92) | 3.14 (2.61)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Lidocaine and Normal Saline Push | Ketorolac and Normal Saline Drip | Lidocaine and Ketorolac
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT02902770/Prot_SAP_000.pdf